CLINICAL TRIAL: NCT01378559
Title: Patient Satisfaction and Complications With the New Titan® One Touch Release (OTR) Penis Prosthesis
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: Titan-2011
Record Dates: First submitted 2011-06-15; First posted 2011-06-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Erectile Dysfunction; Intraoperative Complications; Postoperative Complications
Keywords: Penis prosthesis; Titan; Satisfaction; Complications
MeSH Terms: conditions — Erectile Dysfunction; Intraoperative Complications; Postoperative Complications; Personal Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Penis prosthesis cohort
  Interventions: Other: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire

INTERVENTIONS:
Other: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire — A questionnaire accessing satisfaction with a penis prosthesis

SUMMARY:
The purpose of this study is to assess patient satisfaction with the Titan one touch release penis prosthesis and to register complications with this prosthesis. This will regard the first prostheses inserted at Herlev Hospital/Frederikssund Hospital.

Patient satisfaction will be assessed by mailing out the "Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire" and recording the patient answers. The most important question will be "Overall how satisfied are you with penile prosthesis?".

Complications (including infection, bleeding, and mechanical failure) will be assessed by a patient chart review and confirmed by a brief phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Men who have had a Titan one touch release penis prosthesis implanted at Herlev Hospital.

Exclusion Criteria:

* Inability to read Danish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who have had a Titan one touch release penis prosthesis implanted at Herlev Hospital / Frederikssund Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction assessed by EDITS question 1 | Satisfaction will be assessed when questionnaires are returned - expected avarage 2 months
  Patient satisfaction assesed by the "Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire", Question 1:
  1. Overall how satisfied are you with penile prosthesis? Very satisfied Somewhat satisfied Neither satisfied or dissatisfied Somewhat dissatisfied Very dissatisfied

SECONDARY OUTCOMES:
Complications | At the beginning of study when the chart review is conducted
  Complications may include:
  Bleeding, Infection, Mechanical problems with the device, Erosion, Pain, Penile shortening, Auto inflation, Other complications.
  The number and nature of all complications will be noted. Complications are assessed by patient chart review and a brief phone interview with the patient.
Patient satisfaction assessed by EDITS questions 2-13 | Satisfaction will be assessed when questionnaires are returned - expected avarage 2 months
  "Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire" questions 2-13 include questions about:
  Expectations Continued use of device Ease and frequency of use Confidence Partner satisfaction Erectile function Future surgery Recommendations for others

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sønksen, MD, PhD, Principal Investigator — Herlev Hospital, University of Copenhagen
Locations (1):
- Department of urology, Herlev Hospital, Herlev, Denmark